CLINICAL TRIAL: NCT03132935
Title: Quality Outcomes in Acute Coronary Syndromes Between Telemedically Supported Paramedics and Conventional On-scene Physician Care
Brief Title: Telemedical vs. Conventional Prehospital Care in Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: TEMS-ACS
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Non-STEMI Acute Coronary Syndrome; ST-segment elevation myocardial infarction; Telemedicine
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telemedicine group: Telemedical care of acute coronary syndromes in the prehospital phase. Paramedics were supported by a physician in a tele consultation centre.
  Interventions: Procedure: Telemedical support
- Control group: Conventional on-scene care of acute coronary syndromes by a physician. No telemedicine system was available during this control period.

INTERVENTIONS:
Procedure: Telemedical support — Telemedical support by a physician in a telemedicine centre
  Groups: Telemedicine group

SUMMARY:
Telemedically supported paramedic care of acute coronary syndromes was compared to a historical control period of solely conventional on-scene physician care. Quality outcomes based on current guidelines were researched als well as time requirements in both groups.

DETAILED DESCRIPTION:
Telemedically supported paramedic care of acute coronary syndromes was compared to a historical control period of solely conventional on-scene physician care. Quality outcomes based on current guidelines were researched als well as time requirements in both groups. All data was collected prospectively for quality management purposes and analyzed retrospectively after ethical approval by the local ethics committee.

ELIGIBILITY:
Inclusion Criteria: symptoms of acute coronary syndrome -

Exclusion Criteria: secondary transfers from hospital to hospital, traumatic chest pain

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who called the emergency medical service and the paramedics suspect acute coronary syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | prehospital phase (0.5-2 hours)
  respiratory / circulatory insufficiency, allergic reaction, cardiac arrest

SECONDARY OUTCOMES:
Correct use of Aspirin | prehospital phase (0.5-2 hours)
  Correct use of Aspirin based on current guidelines
Correct use of unfractionated Heparin (UFH) | prehospital phase (0.5-2 hours)
  Correct use of UFH based on current guidelines
Correct use of Morphine | prehospital phase (0.5-2 hours)
  Correct use of Morphine based on current guidelines
Use of 12-lead-ECG | prehospital phase (0.5-2 hours)
  Use of 12-lead-ECG after first medical contact
Correct transport destination | prehospital phase (0.5-2 hours)
  hospital with cath lab in ST-segment elevation myocardial infarction or high-risk Non-STEMI-ACS
Correct use of oxygen | prehospital phase (0.5-2 hours)
  Correct use of Morphine based on current guidelines
Correct use of Glyceroltrinitrate | prehospital phase (0.5-2 hours)
  Correct use of Glyceroltrinitrate based on current guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No